CLINICAL TRIAL: NCT00063128
Title: Safety and Efficacy of Human Insulin Inhalation Powder in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 6944; H7U-MC-IDAI
Record Dates: First submitted 2003-06-20; First posted 2003-06-25 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: insulin
- B (Active Comparator)
  Interventions: Drug: human insulin inhalation powder (HIIP)

INTERVENTIONS:
Drug: insulin — * Administer subcutaneous regular human insulin 30 to 60 minutes before meals, or administer insulin lispro within 15 minutes before meals.
  * Inject into abdomen only.
  Other Names: LY041001
  Arms: A
Drug: human insulin inhalation powder (HIIP) — * Administer HIIP within 15 minutes before meals.
  * Administer doses in one-capsule increments equivalent to approximately 2 IU or 6 IU of subcutaneous insulin.
  * Target treatment goals during the treatment sequence are the same as for patients using preprandial injectable insulin
  Other Names: LY041001
  Arms: B

SUMMARY:
This is a research study of a study drug known as LY041001 or human insulin inhalation powder (HIIP). HIIP is a powder form of insulin made to be inhaled through the mouth and into the lungs using a special handheld device.

ELIGIBILITY:
Inclusion Criteria:

* You are at least 18 years old.
* You have had type 1 diabetes for at least 2 years.
* You are injecting insulin lispro (Humalog), an insulin lispro mixture (Humalog Mixture), regular human insulin mixture (Humulin mixture) before meals using a syringe or injection pen, not an insulin pump.
* If you are female and could become pregnant, you test negative for pregnancy based on blood test at the beginning of the study, do not intend to become pregnant, and agree to use a form of birth control approved by the investigator during the study.
* You have not smoked for at least 1 year, and you agree not to smoke or use smokeless tobacco during the study.

Exclusion Criteria:

* You have used an experimental drug during the last 30 days or have ever taken part in a study of any type of inhaled insulin.
* You have a history of asthma or allergies.
* You have a chronic cough.
* You have had a kidney transplant, are on dialysis, or have poor kidney function.
* You have a history of chest pain, heart attack, or you have a heart condition that limits your physical activity due to discomfort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2003-04; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
test the hypothesis that preprandial HIIP plus insulin glargine is noninferior to preprandial injectable insulin (regular human insulin or insulin lispro) plus insulin glargine with respect to HbA1c | 12 weeks per therapy

SECONDARY OUTCOMES:
compare the pharmacokinetics of test doses of preprandial HIIP and preprandial injectable insulin (regular human insulin or insulin lispro) administered to a subgroup of patients
compare 7-point self-monitored blood glucose profiles (blood glucose measurements before & 2 hours after start of morning, midday, evening meals, and blood glucose measurement at bedtime) for preprandial HIIP and preprandial inject
assess the safety of HIIP using pulmonary function tests, chest x rays, insulin antibody titers, adverse events (AEs), and episodes of hypoglycemia
assess symptoms of diabetes, patient vitality, and patient satisfaction with the diabetes treatments
compare insulin dose requirements (both preprandial and basal insulin [insulin glargine]) of patients administering preprandial HIIP and preprandial injectable insulin (regular human insulin or insulin lispro
assess insulin inhaler reliability
assess patient compliance with the HIIP delivery system Directions for Use (DFU)
assess the impact of practice inhalations on inspiratory flow parameters (peak inspiratory flow rate [IFR] and total inspired volume [TIV]) achieved by patients using the insulin inhaler following training with the DFU

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- United States (25):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Port Richey, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ocala, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pembroke Pines, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jackson, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chesterfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamptom, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flushing, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Hyde Park, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salem, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Federal Way, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Renton, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tacoma, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, West Virginia

REFERENCES:
- [Derived] Hayes RP, Muchmore D, Schmitke J. Effect of inhaled insulin on patient-reported outcomes and treatment preference in patients with type 1 diabetes. Curr Med Res Opin. 2007 Feb;23(2):435-42. doi: 10.1185/030079906X167381. PMID 17288697
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com